CLINICAL TRIAL: NCT02864888
Title: A Controlled, Study of the Effect of Combination Antineoplaston Therapy [Atengenal (A10) and Astugenal (AS2-1)] on the QT/QTc Interval In Subjects With Newly Diagnosed Diffuse, Intrinsic, Brainstem Glioma
Brief Title: Effect of Antineoplaston Therapy on the QT/QTc Interval In Subjects With Diffuse, Intrinsic, Brainstem Glioma
Acronym: DBSG
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BRI-BT-53
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Brain Stem Glioma
Keywords: Diffuse, intrinsic brain stem glioma; QT/QTc interval; Radiation; Antineoplaston therapy
MeSH Terms: interventions — Radiation; antineoplaston A10

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Radiation (Experimental): Study subjects receive a single daily radiation fraction of 180cGy, 5 days a week, for the 2 weeks of the QT/QTc study and for 6 weeks overall to a total radiation dose of 1600 cGy and 5400cGy, respectively.
  Interventions: Radiation: Radiation
- Antineoplaston therapy + Radiation (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 24 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.Study subjects also receive a single daily radiation fraction of 180cGy, 5 days a week, for the 2 weeks of the QT/QTc study and for 6 weeks overall to a total radiation dose of 1600 cGy and 5400cGy, respectively.
  Interventions: Radiation: Radiation; Drug: Atengenal; Drug: Astugenal

INTERVENTIONS:
Radiation: Radiation — Children with a diffuse, intrinsic brain stem glioma will receive radiation.
Drug: Atengenal — Children with a diffuse, intrinsic brain stem glioma will receive Atengenal in combination with Astugenal (Antineoplaston therapy) and radiation
  Other Names: A10
  Arms: Antineoplaston therapy + Radiation
Drug: Astugenal — Children with a diffuse, intrinsic brain stem glioma will receive Astugenal in combination with Atengenal (Antineoplaston therapy) and radiation
  Other Names: AS2-1
  Arms: Antineoplaston therapy + Radiation

SUMMARY:
The primary objective of this protocol study is to investigate the effect of Antineoplaston therapy on the QT/QTc interval in study subjects age 3 to 21 years with newly-diagnosed, diffuse, intrinsic brainstem glioma. This investigation is to be conducted in parallel with a phase 3 efficacy and safety study of combination Antineoplaston therapy + radiation vs. radiation alone (BRI-BT-52).

DETAILED DESCRIPTION:
QT/QTc interval prolongation is investigated during the first two weeks of subject participation in the parallel phase 3 study. The pre-cordial leads and lead II will be utilized to determine QT/QTc prolongation. Descriptive information is provided on changes in T and U wave morphologies. The percentage of subjects in each therapy group who have worsening of the T and U wave morphology is documented. Discrete U waves are excluded from the QT/QTc interval measurement. Except for the pre-therapy ECGs, all ECGs are performed during one ANP therapy infusion daily, that being an afternoon infusion to account for diurnal variation in the QT/QTc interval. The study subject is at rest in the supine position for 30 minutes prior to the ECG study. The baseline QTc is derived from 3 ECGs taken on day 1 during the hour preceding the first Antineoplaston therapy infusion or the first radiation session.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in BRI-BT-52

Exclusion Criteria:

* Not enrolled in BRI-BT-52

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2027-06 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with an Increase in the QTc interval | 6 weeks
  The mean maximum increase in QTc interval, as determined by repeated ECGs, for the Antineoplaston therapy + Radiation study group and the Radiation only study group.

SECONDARY OUTCOMES:
Number of participants with Alterations in T and U Wave Morphology | 6 weeks
  Alterations in T and U wave morphology, as determined by repeated ECGs, for the Antineoplaston therapy + Radiation study group and the Radiation only study group.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burzynski SR, Janicki TJ, Burzynski GS, Marszalek A. The response and survival of children with recurrent diffuse intrinsic pontine glioma based on phase II study of antineoplastons A10 and AS2-1 in patients with brainstem glioma. Childs Nerv Syst. 2014 Dec;30(12):2051-61. doi: 10.1007/s00381-014-2401-z. Epub 2014 Apr 10. PMID 24718705
- [Background] Burzynski SR. Recent clinical trials in diffuse intrinsic brainstem glioma. Cancer Therapy 5:379-390, 2007. Epub 2007 Nov
- [Background] Burzynski SR, Janicki TJ, Weaver RA, Burzynski B. Targeted therapy with antineoplastons A10 and AS2-1 of high-grade, recurrent, and progressive brainstem glioma. Integr Cancer Ther. 2006 Mar;5(1):40-7. doi: 10.1177/1534735405285380. PMID 16484713
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com